CLINICAL TRIAL: NCT00237445
Title: A Multinational, Multicenter, Randomized, Double-blind, Study in Areas of High Pneumococcal Resistance Comparing the Clinical Efficacy and Health Outcomes of Outpatients With Mild to Moderate Community-Acquired Pneumonia (CAP) Treated With Either Ketek® Telithromycin Once Daily for 7 Days, or Zithromax® Azithromycin Once Daily for 5 Days
Brief Title: Study Comparing the Clinical Efficacy and Health Outcomes of Outpatients With Mild to Moderate Community-Acquired Pneumonia (CAP) Treated With Either Telithromycin Once Daily for 7 Days, or Azithromycin Once Daily for 5 Days
Acronym: COBRA II
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR3647A_4027
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — telithromycin; Azithromycin

INTERVENTIONS:
Drug: telithromycin
Drug: azithromycin

SUMMARY:
A multinational, multicenter, randomized, double-blind, study in areas of high pneumococcal resistance comparing the clinical efficacy and health outcomes of outpatients with mild to moderate Community-Acquired Pneumonia (CAP) treated with either telithromycin once daily for 7 days, or azithromycin once daily for 5 days

ELIGIBILITY:
Inclusion Criteria:

Male or female outpatients aged 20 or greater.

* Subjects with a positive Binax NOW S. pneumoniae Urinary Antigen Test and/or positive gram stain for diplococci.
* Subjects with ≤ 7 days of signs and symptoms of CAP.
* Subjects with chest x-ray findings that support a diagnosis of acute pneumonia with presence of a new infiltrate. For subjects with history of chronic obstructive pulmonary disease (COPD), a comparison to previous chest x-ray report is required to confirm the finding of new infiltrates.

Subjects with diagnosis of acute mild to moderate CAP based on at least one of the following:

* fever (oral >37.5°C/99.5°F or axillary >37.4°C/99.4°F or rectal >38.5°C/101.5°F) or
* elevated total peripheral white blood cell count >10,000/mm3 or >15% immature neutrophils (bands), regardless of total peripheral white count and
* new and sudden onset (equal or less than 48 hours) of at least two of the following signs or symptoms:

  * cough
  * dyspnea or tachypnea (particularly if progressive in nature)
  * pleuritic chest pain
  * purulent sputum production or change in sputum character
  * auscultatory findings (such as rales and/or evidence of pulmonary consolidation)

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study.

  * Subjects with CAP requiring hospitalization.
  * Subjects with signs and symptoms of severe CAP lasting greater than 7 days.
  * Subjects requiring parenteral antibiotic treatment.
  * Subjects discharged from hospital within the 10 days before study entry.
  * Subjects with visible/gross aspiration pneumonia.
  * Subjects with any concomitant pulmonary disease, condition or complication that could confound the interpretation or evaluation of drug efficacy or safety, including:
* severe bronchiectasis, cystic fibrosis or suspected active pulmonary tuberculosis
* suspected acute pulmonary embolism
* emphysema, lung abscess, extra pulmonary extension (e.g., meningitis, septic arthritis, endocarditis)
* known bronchial obstruction or a history of postobstructive pneumonia.

  * Subjects with neoplastic lung disease (lung cancer) or another malignancy metastatic to the lungs, and/or requiring chemotherapeutic interventions for this or other neoplasms.
  * Subjects with infection requiring administration of other systemic antimicrobial agents.
  * Subjects with progressively fatal disease; life expectancy ≤3 months.
  * Subjects with myasthenia gravis.
  * Subjects with any concomitant condition, including severe and/or uncontrolled cardiovascular, neurologic, endocrine, or other severe and/or uncontrolled major systemic disease that make implementation of the protocol or interpretation of the study results difficult.
  * Immunocompromised subjects, such as:
* known HIV subjects with CD4+ T-lymphocyte count dated less than 3 months <200/mm3 and /or HIV subjects treated with isoniazide or clarithromycin as prophylaxis
* neutropenia (<1500 neutrophils/mm3) not attributable to the acute infectious disease
* metastatic or hematological malignancy
* splenectomy or known hyposplenia or asplenia
* chronic corticosteroid therapy.

  * Subjects with a history of congenital or a family history of long QT syndrome (if not excluded by previous ECG) and subjects with known acquired QT interval prolongation
  * Known severe impaired renal function as shown by creatinine clearance < 30 ml/min either measured or estimated with Cockroft formula.
  * Subjects who have received more than 24 hours of effective treatment with other antibiotics, within the 7 days prior to enrollment in the study.
  * Subjects with a known or suspected hypersensitivity to, or a known or suspected serious adverse reaction to telithromycin or any macrolide antibiotic.
  * Subjects who will require on-study treatment with medications known to have potential drug interactions, including ergot alkaloids derivatives, terfenadine, astemizole, cisapride, pimozide, simvastatin, atorvastatin and lovastatin (see Section 6.2).
  * Subjects who have received any investigational drug within 1 month prior to study entry or such treatment is planned for during the study period.
  * Subjects who are pregnant or breast-feeding.
  * Subjects with recent drug or alcohol abuse.Subjects with a mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
  * Subject is the investigator or any subinvestigator, research assistance, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
  * Subjects already enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Evaluate clinical cure rates of telithromycin over azithromycin for treating adult outpatients with mild to moderate community-acquired pneumonia (CAP) in high pneumococcal bacterial resistance areas, at the test of cure visit (Days 17-21).

SECONDARY OUTCOMES:
To compare the effect of telithromycin versus azithromycin on clinical efficacy in CAP adult outpatients at the end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States